CLINICAL TRIAL: NCT02385721
Title: A Prospective, Observational, Post-Authorization Long-term Safety Surveillance on Antihypertensive Treatment With Kanarb® (Fimasartan) During 1 Year Among 20 and Older Diagnosed With Essential Hypertension
Brief Title: Post-Authorization Long-term Safety Surveillance on Antihypertensive Treatment With Kanarb® (Fimasartan)
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-FMS-PASS-401
Record Dates: First submitted 2015-03-03; First posted 2015-03-11 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Essential Hypertension
Keywords: Hypertension; Fimasartan
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluated the incidence and characteristics of adverse events during the treatment for Kanarb tablet.

DETAILED DESCRIPTION:
This study is designed to evaluate the incidence and characteristics (profile, relationship to the study drug, severity, and outcome) of adverse events (AEs) observed during 1-year treatment with Kanarb tablet® (fimasartan)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with essential hypertension
2. Taking Kanarb tablet® (fimasartan) as prescribed previously (within 1 month) or newly
3. Male and female adults aged 20 years or older
4. Voluntarily provided a written consent to participate in the study

Exclusion Criteria:

1. Patients with hypersensitivity to this drug or the ingredients of this drug
2. Pregnant or breast-feeding women
3. Patients on renal dialysis
4. Patients with moderate to severe hepatic impairment
5. Patients with biliary atresia
6. Genetic disorders such as galactose intolerance, lapp lactase deficiency, or glucose-galactose malabsorption
7. Patients considered inappropriate for taking Kanarb tablet® (fimasartan) by investigator
8. Clinically significant abnormal liver function (AST, ALT ≥2 x upper limit of normal (ULN); TB ≥1.5 ULN)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertension Patients
Sampling Method: Probability Sample
Enrollment: 601 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myung Sook Hong, Study Director — Boryung Pharmaceutical Co., Ltd
Locations (1):
- Yoon Jun Kim, Seoul, South Korea

REFERENCES:
- [Derived] Oh GC, Joo KW, Kim MA, Choi DJ, Kim YJ, Lee HY. Long-Term Safety of a Novel Angiotensin Receptor Blocker, Fimasartan, According to the Absence or Presence of Underlying Liver Disease in Korean Hypertensive Patients: A Prospective, 12-Month, Observational Study. Drug Des Devel Ther. 2020 Apr 3;14:1341-1349. doi: 10.2147/DDDT.S233174. eCollection 2020. PMID 32308367

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety Set: Patients with essential hypertension who received Kanarb tablet® (fimasartan)
Period: Overall Study
Arm/Group | Safety Set
Started | 601
Completed | 371
Not Completed | 230

BASELINE CHARACTERISTICS:
Arm/Group | Safety Set
Number analyzed (Participants) | 601
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.65 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267
  Male | 334
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.34 (3.31)
Duration of Hypertension [Mean (Standard Deviation); unit: years] | 6.47 (8.52)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing AEs or ADRs
Description: Number of participants experiencing AEs (or ADRs) during the study
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Set
Number analyzed (Participants) | 601
Participants
  AE | 184
  ADR | 59

2. Secondary Outcome: Treatment Persistence Rate of Fimasartan
Description: Treatment persistence rate of Kanarb tablet® (fimasartan) until the end of 1-year study
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Set
Number analyzed (Participants) | 601
Participants
  Study completion | 371
  Study withdrawn | 230

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Safety Set
All-Cause Mortality (participants affected / at risk) | 0/601
Serious Adverse Events (participants affected / at risk) | 33/601
Other Adverse Events (participants affected / at risk) | 59/601
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Set (N=601)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Azotaemia (Renal and urinary disorders) | 1 (1)
Glomerulonephritis membranous (Renal and urinary disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Infective spondylitis (Infections and infestations) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Set (N=601)
Dizziness (Nervous system disorders) | 14 (15)
Headache (Nervous system disorders) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4)
Blood pressure increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood pressure decreased (Investigations) | 5 (5)
Liver function test abnormal (Investigations) | 1 (1)
Liver function test increased (Investigations) | 1 (1)
Dyspepsi (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 3 (3)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 8 (8)
Hot flush (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT02385721/Prot_SAP_000.pdf